CLINICAL TRIAL: NCT06877988
Title: Artificial Intelligence (AI) - Assisted Visual Impairment Screening Model: Community-based Implementation and Evaluation of Performance, Feasibility and Costs.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Eye Research Institute (Other)
Collaborators: Institute of High Performance Computing (IHPC), A*STAR Research Institutes (Unknown); National University Polyclinics, Singapore (Other)
Responsible Party: Principal Investigator, Tham Yih Chung, Principal Investigator, Singapore Eye Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2024/2297
Record Dates: First submitted 2025-03-07; First posted 2025-03-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Visual Impairment
Keywords: Visual impairment; Community Screening; Randomized Controlled Trial (RCT); Artificial Intelligence (AI)
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AI-assisted (Experimental): Participants will undergo visual impairment screening using AVIRI model (AI for Disease-related Visual Impairment Screening Using Retinal Imaging). This intervention involves automated fundus image analysis through artificial intelligence to screen and identify individuals with high probability of visual impairment.
  Interventions: Device: AI
- Traditional (No Intervention): Participants will receive visual impairment screening using the traditional screening model, which involves optometrists performing initial assessments, followed by referral decisions based on manual fundus image evaluation.

INTERVENTIONS:
Device: AI — Retinal photography-based deep learning algorithm for detection of disease-related visual impairment cases
  Other Names: AVIRI (AI for Disease-related Visual Impairment Screening Using Retinal Imaging)
  Arms: AI-assisted

SUMMARY:
The goal of this observational study is to evaluate the performance, operational efficiency, acceptability, feasibility, and cost-effectiveness of an AI-assisted screening model for visual impairment in a community setting. The main questions it aims to answer are:

* Can the AI-assisted screening model improve screening and referral accuracy compared to the current traditional screening approach?
* Does the AI-assisted model enhance operational efficiency and reduce healthcare costs in a community setting?

Researchers will compare the AI-assisted model with the current traditional screening approach to assess its impact on screening accuracy, operational efficiency, and cost-effectiveness.

Participants will:

* Undergo vision screening using either the AI-assisted model or the traditional model.
* Provide feedback on the acceptability of the screening approach.
* Contribute to evaluating the feasibility and costs associated with each screening method.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 50 years old and above.

Exclusion Criteria:

* Individuals aged below 50 years old.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Performance of AVIRI on the detection of visual impairment | through study completion, an average 1 year
  The primary outcome is the detection performance for VI (refractive error-related and disease-related VI) and the rate of correct referral, with reference to the expert panels' diagnosis . To assess whether the new AI-assisted model has better referral accuracy than the current traditional model, the accuracy, AUC values, sensitivity, specificity and other performance metrics of the two models will be calculated and compared.

SECONDARY OUTCOMES:
Operational efficiency | through study completion, an average 1 year
  Evaluation includes (i) average screening time per patient and (ii) average number of patients screened per session.
Patient acceptability | through study completion, an average 1 year
  Patient Acceptability is assessed via a 6-item questionnaire (4-point Likert scale: 'Satisfaction' or 'Likelihood') administered by trained coordinators.
Perceptions of feasibility | through study completion, an average 1 year
  Perceptions of feasibility is evaluated through at least two focus groups with optometrists and one with service providers will be conducted, guided by the Consolidated Framework for Implementation Research (CFIR). Discussions will explore barriers and facilitators influencing the AI screening model's adoption. Data will be inductively and deductively coded by two researchers using CFIR constructs; discrepancies resolved through consensus or a third researcher.
Cost savings of implementing the AI-assisted screening model | through study completion, an average 1 year
  Researchers will quantify the incremental cost savings of implementing the AI-assisted screening model over the PSS model using an Activity Based Costing (ABC) approach that quantifies all non-sunk costs (including labor, materials and supplies, and amortized technology and space utility/ rental costs) required to conduct each assessment stratified by key activities of each screening model (e.g., conduct screening examinations, operationalize the AVIRI algorithm, on-site generation of test results etc.). Fixed costs will be amortized over the inputs' expected useful life (i.e. involved fixed assets' life expectancy). For the cost of clinical assessments, researchers will use non-subsidized bill sizes as these are expected to approximate actual costs.

CONTACTS AND LOCATIONS:
Locations (1):
- Pioneer Polyclinic, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided